CLINICAL TRIAL: NCT06325163
Title: Accuracy of Artificial Intelligence Technology in Detecting Number of Root Canals in Human Mandibular First Molars Obturated and Indicated for Retreatment: Diagnostic Accuracy Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Albaraa Samir Abdelrwab Alkady, Principle investigator, Misr International University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MIU-IRB-2223-219
Record Dates: First submitted 2023-12-26; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Missed Canals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single arm consisting of 3 stages (Experimental): This study will include 3 stages:
  1. CBCT examination stage: In this stage, CBCT scanning will be done and examined by by 2 blinded endodontists and the number of canals identified will be recorded
  2. Clinical Stage: This is a clinical stage where patients will be randomly distributed upon 6 Practitioners using randomization software (Microsoft Office Excel). Practitioners will then proceed with the pretreatment procedures under dental operating microscope
  3. Artificial intelligence stage: The carrying out of this stage will be solely undertaken by the principal investigator. The CBCT images will be uploaded to convolutional neural network software (CNN) that uses a deep learning algorithm and CBCT segmentation. The software will then record the number of canals it found
  Interventions: Diagnostic Test: CBCT; Diagnostic Test: clinical examination under dental operating microscope; Diagnostic Test: canal detection AI software (diagnocat)

INTERVENTIONS:
Diagnostic Test: CBCT — Mandibular molar indicated for retreatment will be scanned using limited field of view CBCT to examine the number of canals
Diagnostic Test: clinical examination under dental operating microscope — the number of canals will be examined by an a randomly assigned operator following gutta percha removal under dental operating microscope
Diagnostic Test: canal detection AI software (diagnocat) — software used to analyze CBCT images and report the number of canals

SUMMARY:
evaluate the accuracy of new AI technology for detecting root canals in mandibular first molars retreatment cases in comparison to dentist clinical access cavity and CBCT imaging.

DETAILED DESCRIPTION:
evaluate the accuracy of new AI technology for detecting root canals in mandibular first molars retreatment cases in comparison to dentist clinical access cavity and CBCT imaging.

1. CBCT exmanation stage: In this stage, CBCT scanning was done using Soredex Cranex 3D Dental Imaging System, FINLAND, with the following parameters ((XS FOV dimensions 61 x 41 mm (HxD)) (XS FOV High resolution 90 kV / 4 - 12.5 mA / 6.1 s)).

   The samples will be randomized using randomization software (Microsoft Office Excel, USA) and will be assigned randomly to 2 endodontists who are unaware of the findings of stage 2. After interpreting and segmenting the CBCT scans in DICOM Format using OnDemand software (USA), the number of canals identified will be recorded on a pre-established information guide.

   The samples are coded based on the patient's file number, and the codes were undisclosed so that the CBCT examiners could not identify the samples. All images were interpreted from the axial section in the analysis of the tomographic sections, the number of canals are identified by the corresponding radiolucent orifices, regardless of their location along the root
2. Clinical Stage: This is a clinical stage where the thirty-five patients, as predetermined by power analysis, will be randomly distributed upon 6 Practitioners using randomization software (Microsoft Office Excel). Practitioners will then proceed in access formation under dental operating microscope, (Leica M320D using magnification 16X, using fully integrated 4K camera).

   Access will be done using TR13 diamond stone (Mani, Japan) to remove caries and restorations.

   Troughing will be done using ultrasonic tip (NSK E4 and E15D) power 3W.

   Irrigation will be done using NAOCL (JK Dental Vision sodium hypochlorite, Egypt) with a concentration of 2.5%.

   Gutta percha will be removed from the canal using M-pro rotary files:

   At first orifice opener will be used to remove the coronal gutta percha then used the yellow file tapered 4% then confirm the working length by apex locator, after that using taper file 25 to remove the remaining gutta percha.

   DG16 endodontic probe (Dentsply Sirona, Germany) will be used to locate canal orifices.

   Upon confirmation by clinic PHD supervisors, the number of orifices found will be recorded on a pre-formed information guide, in one visit per patient. Access cavity will be aided by Leica M320D DOM
3. Artificial intelligence stage: The carrying out of this stage will be solely undertaken by the principal investigator. The CBCT images will be uploaded to convolutional neural network software (CNN) that uses a deep learning algorithm and CBCT segmentation. The software will then record the number of canals it found

The software utilized employs deep convolutional neural networks (CNNs) with a specific U-net inspired structure. The complete CBCT scan is uploaded onto the software, where all collected images are analyzed and each tooth in the 3D scan is precisely located and assessed. The software uses pattern recognition and statistical predictions to segment numerous slices of each tooth and determine the condition or pathosis present. This is achieved by analyzing previously fed photos that were used to train the software

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* Patients aged 18 to 40 years
* Repairable permanent first molars in the lower jaw, with a closed apex, which required non-surgical retreatment.
* One or more of the following signs and symptoms: Spontaneous pain, Pain on biting, Sinus tract, Radiolucency related to one or more roots.

Exclusion Criteria:

* Patients with lower first molars which are deemed non restorable, or have large perforations, external resorption, or vertical root fracture,
* Pregnant women
* Immunocompromised patients.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Number of canals | The day of the procedure
  the numbers of canals in mandibular molars indicated for retreatment will be measured using CBCT, clinical under dental operating microscope, and using AI software

SECONDARY OUTCOMES:
linear morphological variations in failed cases | Following the CBCT stage, an average of one week
  This outcome will measure I)Inter orifice distance II)Canal configuration. III)Width of the root, in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International University, Cairo, Egypt